CLINICAL TRIAL: NCT05121948
Title: A Multicenter, Open-label, Phase 1a/b Study of HC-7366 in Subjects With Advanced Solid Tumors
Brief Title: A Study of HC-7366 to Establish the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: HiberCell, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HC366-FCP2111
Record Dates: First submitted 2021-11-05; First posted 2021-11-16 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Colo-rectal Cancer; Non Small Cell Lung Cancer; Transitional Cell Carcinoma of the Bladder; Other Solid Tumors; Clear Cell Renal Cell Carcinoma
Keywords: SCCHN; CRC; NSCLC; TCC; Phase 1; First in human; HC-7366; ccRCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 1a Cohort 1 - 10 mg (Experimental): 10 mg capsules of HC-7366 administered orally once a day in the fasting state with water at least 1 hour before food or at least 2 hours after food of each 3-week treatment cycle
  Interventions: Drug: HC-7366
- Phase 1a Cohort 2 - 20 mg (Experimental): 20 mg capsules of HC-7366 administered orally once a day in the fasting state with water at least 1 hour before food or at least 2 hours after food of each 3-week treatment cycle
  Interventions: Drug: HC-7366
- Phase 1a Cohort 3 - 40 mg (Experimental): 40 mg capsules of HC-7366 administered orally once a day in the fasting state with water at least 1 hour before food or at least 2 hours after food of each 3-week treatment cycle
  Interventions: Drug: HC-7366
- Phase 1a Cohort 4 - 75 mg (Experimental): 75 mg capsules of HC-7366 administered orally once a day in the fasting state with water at least 1 hour before food or at least 2 hours after food of each 3-week treatment cycle
  Interventions: Drug: HC-7366
- Phase 1a Cohort 5 - 125 mg (Experimental): 125 mg capsules of HC-7366 administered orally once a day in the fasting state with water at least 1 hour before food or at least 2 hours after food of each 3-week treatment cycle
  Interventions: Drug: HC-7366
- Phase 1a Cohort 6 - 150 mg (Experimental): 150 mg capsules of HC-7366 administered orally once a day in the fasting state with water at least 1 hour before food or at least 2 hours after food of each 3-week treatment cycle
  Interventions: Drug: HC-7366
- Phase 1b Cohort 7 - Dose 1 Chosen for Expansion (Experimental): XX mg capsules of HC-7366 administered orally once a day in the fasting state with water at least 1 hour before food or at least 2 hours after food of each 3-week treatment cycle
  Interventions: Drug: HC-7366
- Phase 1b Cohort 8 - Dose 2 Chosen for Expansion (Experimental): XX mg capsules of HC-7366 administered orally once a day in the fasting state with water at least 1 hour before food or at least 2 hours after food of each 3-week treatment cycle
  Interventions: Drug: HC-7366

INTERVENTIONS:
Drug: HC-7366 — HC-7366 drug product is an immediate release capsule formulation of HC-7366 potassium salt monohydrate (HC-7366-K) in a hard gelatin capsule for oral administration. Each capsule contains HC-7366-K monohydrate (the active ingredient), lactose monohydrate, microcrystalline cellulose, croscarmellose sodium, colloidal silicon dioxide, and magnesium stearate. Capsules are supplied in 3 strengths: 10, 25, and 100 mg HC-7366 free acid equivalent.

SUMMARY:
This is a first in human, multicenter, open label, Phase 1a and 1b dose-escalation and dose-expansion study to establish the maximum tolerated dose, recommended Phase 2 dose, and evaluate the safety and tolerability of QD oral dosing of HC 7366 in a dose escalating fashion in subjects with advanced solid tumors. Up to 40 subjects will be enrolled into the Phase 1a dose-escalation part of the study. The study will be conducted in the United States at approximately 7 to 10 sites. Every effort will be made to ensure approximately 50% of all subjects enrolled into Phase 1a of this study are subjects with the tumors of special interest including squamous cell carcinoma of the head and neck, colorectal cancer, non-small cell lung cancer, and transitional cell carcinoma of the bladder. Subjects with other solid tumor types are also eligible provided study selection criteria are met and they do not exceed 50% of all enrolled subjects. All subjects in Phase 1b will enroll with clear cell renal cell carcinoma. The Phase 1a study will follow a traditional 3+3 design. The starting dose level will be 10 mg QD, escalating to 20, 40, 75, 125, and 150 mg QD as safety allows. All doses are to be administered in the fasting state with water at least 1 hour before food or at least 2 hours after food. The Phase 1b dose-expansion will be at a single dose level of 75 mg based on the safety, tolerability, PK/PD results from Phase 1a to obtain additional safety and preliminary efficacy information. At the discretion of the safety monitoring committee and sponsor, the cohort may be expanded to enroll additional patients and/ or 1-2 additional cohorts will be opened. Up to 30 subjects may be enrolled in the Phase 1b portion of the study at the 75 mg dose. Replacement patients will be enrolled if necessary. Subjects will be dosed until unacceptable toxicity, disease progression per immune-related Response Evaluation Criteria in Solid Tumors, discontinuation of treatment for other protocol allowed reason (eg, subject refusal), any other administrative reasons, or after 2 years of treatment, whichever occurs first. For scheduling purposes, dosing in Phase 1a and 1b will occur in 3 week cycles and computed tomography scans will be conducted once every 6 weeks from Cycle 1/Day 1, with the first postbaseline scan after 6 weeks of dosing (precycle 3) until confirmed disease progression, death, start of new anticancer therapy, withdrawal of consent, or end of study, whichever occurs first.

DETAILED DESCRIPTION:
Subjects of Phase 1a and 1b are to spend Cycle 1/Day 1 (C1D1) in the clinic followed by an optional overnight stay for safety monitoring and PK sampling. Subjects will be hospitalized (optional) for administration of the first 2 doses: C1D1 and Cycle 1/Day 2 (C1D2). After the initial optional hospital stay at the start of study, subjects will be seen in the outpatient clinic on Days 8, 15, and 21 of Cycle 1 and thereafter, on the first day of each cycle for physical and laboratory assessments, adverse event (AE) and dosing compliance monitoring, and PK C3-C6; the End of Treatment visit will also be in-person in the outpatient clinic. An overnight stay for Cycle 1/Day 21 (C1D21) to C2D1 is also optional. Subjects will be allowed to go home after having a 12-hour PK sample draw in the clinic and will be asked to return to the clinic on C1D2 (for a safety check with a PK sample draw and an electrocardiogram (ECG) prior to dosing.

Subjects of Phase 1a who discontinue before the first postbaseline CT scan for reasons other than disease progression, a treatment-related AE, or dose limiting toxicity (DLT) prior to completion of the DLT evaluation period will be replaced to ensure an adequate safety assessment at each dose level. Subjects of Phase 1b who discontinue before the first postbaseline CT scan for reasons other than disease progression, or a treatment-related AE will be replaced and will be censored for efficacy; however, enrollment will continue to include enough subjects at each dose level in order to complete safety and efficacy assessments of that dose level.

Each subject in Phase 1a and 1b will be treated for a maximum of 2 years and followed for a maximum of 2 years.

Six dose-escalation levels are planned for subjects in the Phase 1a part of the study. Dose escalation will follow a traditional 3+3 design. A minimum of 3 subjects will be enrolled in each cohort sequentially, with expansion to 6 subjects in each cohort as needed to determine the DLT. For each cohort, the first subject is a sentinel subject. Sentinel subjects will be dosed and followed for 4 days to assess safety and tolerability. If deemed safe and well tolerated, the remainder of the cohort (N=2) will be enrolled. If none of the first 3 subjects in a cohort experiences a study treatment related DLT during the first 21 days (DLT evaluation period), the next cohort may be enrolled. Before applying the dose escalation rules, 3 subjects in a given dose level must have received a minimum of 75% of the planned dose and have been evaluated for toxicity, unless one or more subjects experiences a DLT within the first 21 days. If the first 3 DLT-evaluable subjects within a cohort experience no DLTs during the DLT-evaluation period, the next cohort may enroll. In the case a subject does not receive a minimum of 75% of the planned dose, for any reason other than a DLT (ie, lost to follow-up), the subject may be replaced. DLT's will be reviewed by the Safety Monitoring Committee (SMC) when the planned number of subjects of Phase 1a part of the study complete their DLT observation period using the dose-escalation rules. If the MTD is not reached even at the maximum dose level (150 mg QD is well tolerated), a higher dose level may be evaluated based on the SMC recommendations after a comprehensive review of the safety, PK, and efficacy data generated from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a signed an informed consent form prior to any study specific procedures or treatment
2. Be ≥18 years of age (male or female) at the time of consent
3. Phase 1a:

   Have 1 of the following tumor types with qualifying characteristics, and have received at least 1 and no more than 5 prior lines of therapy for metastatic (stage IV) disease:
   1. SCCHN
   2. CRC
   3. NSCLC
   4. TCC
   5. Other solid tumors (eg, carcinoma of unknown primary) with the exception of rapidly progressing neoplasms (eg, pancreatic cancer, glioblastoma, hepatocellular carcinoma). Note: Subjects do not need to have progressed through all possible available therapies with known clinical benefit for their respective cancers to participate in this study. Note: Subjects with SCCHN, CRC, NSCLC, and TCC are a priority and should constitute as a whole, at least 50% of the enrolled population. Enrollment of all others will be capped when reaching a combined 50%, in order to maintain 18 slots for subjects with SCCHN, CRC, NSCLC, and TCC.

   Phase 1b:

   Have renal cell carcinoma with respective qualifying characteristics:
   1. Histological or cytological proof of component (any percentage) of clear cell RCC, excluding subjects that have any component of collecting duct or medullary histology are eligible
   2. Subjects with residual, but well-controlled endocrinopathy (eg, hypothyroidism) are eligible
   3. Subjects with metastatic or locally advanced unresectable RCC Note: Prior nephrectomy is not mandatory.
   4. Subjects with progressive disease after receipt of at least 2 and no more than 5 prior lines of therapy for metastatic (stage IV) disease, including but not limited to VEGF-directed tyrosine kinase inhibitors (TKIs), high-dose IL-2 , immune checkpoint inhibitors, mTOR inhibitors, or belzutifan, alone or in combination. Note: A line of therapy is considered complete once the patient has progressed following such treatment. If a treatment regimen is changed before disease progression due to toxicity, for example, this is still considered part of the same line of therapy. In addition, maintenance therapy [that is, therapy with a different drug or drugs given to conserve an existing response or stable disease before disease progression] is not considered an additional line of therapy.
4. Have at least 1 radiologically measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 defined as a lesion that is at least 10 mm in longest diameter or lymph node that is at least 15 mm in short axis imaged by CT scan or magnetic resonance imaging and obtained by imaging within 28 days prior to study treatment. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
5. Have resolution of all previous treatment related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (≤Grade 2) and alopecia. If the subject received major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or complications from the intervention
6. If subjects were previously treated with immune checkpoint inhibitors, at least 4 weeks must have elapsed since the last dose, and they must have recovered from toxicities as mentioned in above Criterion #5
7. Subjects must have at least one biopsiable lesion at baseline. Biopsies in this clinical study will conform to American Society of Clinical Oncology's Ethical Framework for Including Research Biopsies in Oncology Clinical Trials. Provided there are suitable and accessible lesions, no biopsy contraindications, minimal risk of complications and a positive informed decision, subjects are willing to provide fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality, for assessment of biomarker status. Two biopsies will be necessary: at baseline (within 15 days prior to study Day 1) and at the time of the first response assessment CT scan at Cycle 3/Day 1 (+7 days). Newly obtained biopsy specimens are preferred to archived samples and formalin fixed, paraffin embedded block specimens are preferred to slides. Biopsies should not be taken from target lesions
8. Have Eastern Cooperative Oncology Group performance status of 0 or 1 and sustained between screening and initiation of dosing on Day 1
9. Have no swallowing difficulties that would prevent compliance with oral dosing
10. Have not experienced >10% body weight loss in the previous 4 weeks
11. Have a serum albumin level >3 g/dL
12. Have life expectancy of 3 months or greater as determined by the treating physician
13. Have adequate organ function on Day 1, as defined by meeting all of the following criteria:

    1. Total bilirubin ≤1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5 x ULN
    2. Aspartate aminotransferase and alanine aminotransferase ≤2.5 × ULN or ≤5 × ULN for subjects with known hepatic metastases
14. Have adequate renal function on Day 1, as defined by creatinine ≤1.5 × ULN and creatinine clearance ≥60 mL/min, as per the below Cockcroft Gault formula
15. Have adequate hematologic function on Day 1, as defined by meeting all of the following criteria:

    1. Hemoglobin ≥9 g/dL (uncorrected by red blood cell transfusion or erythropoietin support)
    2. Absolute neutrophil count ≥1.5 × 109/L
    3. Platelet count ≥100 × 109/L
16. Have adequate coagulation function on Day 1, as defined by either of the following criteria:

    1. International normalized ratio (INR) <1.5 × ULN OR for subjects receiving warfarin or low molecular weight heparin, the subject must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these subjects may exceed 1.5 × ULN if that is the goal of anticoagulant therapy
    2. Activated partial thromboplastin time <1.5 × ULN unless subject is receiving anticoagulant therapy, provided prothrombin time or partial thromboplastin time is within therapeutic range of intended use of anticoagulants
17. Have normal or adequately controlled pan-endocrine function (pituitary, adrenal, thyroid, pancreatic, gonadal). Subjects on hormonal supplementation must be stable at their treatment doses
18. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
19. Female subjects of childbearing potential must be willing to use an adequate form of contraception from the signing of the ICF until 90 days after the last dose of study medication
20. Female subjects must agree not to breastfeed and not to donate ova starting at screening and throughout the study treatment, and for 90 days after the final administration of study drug
21. Male subjects with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or for the time their partner is breastfeeding throughout the study treatment and for 90 days after the final administration of study drug
22. Male subjects must not donate sperm during the treatment period and for at least 90 days after the final administration of the study drug
23. Male subjects with female partner(s) of child bearing potential must agree to use a condom with spermicide during the treatment period and for at least 90 days after the final administration of the study drug
24. Be willing and have the ability to comply with scheduled visits (including geographical proximity), treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of study treatment or who has not recovered from adverse reactions due to a previously administered agent or major surgery
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
3. Has a diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor
4. Has known history of active tuberculosis
5. Has known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
6. Has known active hepatitis B (eg, hepatitis B surface antigen reactive) or hepatitis C (eg, hepatitis C virus ribonucleic acid [RNA] [qualitative]) infection
7. Has been diagnosed with any infectious process that would, in the opinion of the investigator, interfere with study participation, especially regarding site-specific testing and isolation requirements. This applies to viral infections including, but not limited to, severe acute respiratory syndrome coronavirus (SARS-CoV-2) infection
8. Has a history of clinically severe autoimmune disease, or history of organ transplant
9. Has a history of retinitis or photosensitive skin disorders including (but not limited to) erythema multiforme, atopic eczema, psoriasis, viral exanthemata, pemphigus, and dermatitis herpetiformis
10. Has known additional malignancy that is progressing or required active treatment within the previous 5 years. Exceptions include basal cell carcinoma or squamous cell carcinoma of the skin that has undergone potentially curative therapy, superficial bladder cancer, or in situ cervical cancer. Subjects with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease free for at least 5 years
11. Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of disease progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using systemic steroids for at least 7 days prior to study treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
12. Has a history of interstitial lung disease, pneumonitis within 12 months prior to screening, or current pneumonitis
13. Has an active infection requiring systemic therapy
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
15. Has a clinically significant cardiovascular disease such as unstable angina, myocardial infarction, or acute coronary syndrome, symptomatic or uncontrolled arrhythmia, congestive heart failure, baseline electrocardiogram (ECG) abnormalities, including, but not limited to, QTc prolongation (as calculated using Fridericia formula) to greater than 450 ms for males or to greater than 470 ms for females, or any Class III or IV cardiac disease as defined by the New York Heart Association Functional Classification
16. Has overt or latent disorders of the exocrine pancreas (such as acute or chronic pancreatitis of any etiology) or chronic (including autoimmune) gastrointestinal disorders such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, lupus, scleroderma, Sjogren's syndrome, and polyarteritis nodosa
17. Has a known psychiatric or substance abuse disorder(s) that would interfere with informed consent or cooperation with the requirements of the study
18. Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through 90 days after the final administration of the study drug
19. Is a first degree relative of the investigator, staff, or study sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Determination of MTD of HC-7366 | Within 18 months of last patient enrolled
  When orally administered once daily in a dose escalating fashion in subjects with selected, advanced solid tumors
Determination of Recommended Phase 2 dose of HC-7366 | Within 18 months of last patient enrolled
  When orally administered once daily in a dose escalating fashion in subjects with selected, advanced solid tumors
Occurrence of dose-limiting toxicities (DLTs) | Within 18 months of last patient enrolled
Incidence and severity of treatment-emergent adverse events (TEAEs) and treatment related TEAEs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 5.0 | Within 18 months of last patient enrolled
Incidence of TEAEs leading to premature discontinuation | Within 18 months of last patient enrolled
Incidence of laboratory abnormalities, based on NCI CTCAE grades of hematology, serum chemistry, and urinalysis test results | Within 18 months of last patient enrolled
Incidence of abnormalities observed in 12 lead ECG parameters | Within 18 months of last patient enrolled
Incidence of abnormalities observed in vital signs measurements | Within 18 months of last patient enrolled

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from time 0 until last measurable concentration (AUC 0-last) | Within 24 months of last patient enrolled
Area under the plasma concentration versus time curve from time 0 to 24 hours postdose (AUC 0-24) | Within 24 months of last patient enrolled
Area under the plasma concentration versus time curve from time 0 extrapolated to infinity (AUC 0-∞) | Within 24 months of last patient enrolled
Area under the plasma concentration versus time curve over a dosing interval (AUC 0-t) | Within 24 months of last patient enrolled
Peak plasma concentration (Cmax) | Within 24 months of last patient enrolled
Time of the maximum observed plasma concentration (tmax) | Within 24 months of last patient enrolled
Apparent total clearance (CL/F) of plasma concentration | Within 24 months of last patient enrolled
Apparent volume of distribution during the terminal phase (Vz/F) of plasma concentration | Within 24 months of last patient enrolled
Apparent terminal elimination half life (t1/2) of plasma concentration | Within 24 months of last patient enrolled
Accumulation ratio based on AUC 0-t (ARAUC) of plasma concentration | Within 24 months of last patient enrolled
Linearity ratio (LR) of plasma concentration | Within 24 months of last patient enrolled
Overall response rate (ORR) to HC-7366 using iRECIST | Within 24 months of last patient enrolled
Duration of response (DOR) to HC-7366 using iRECIST | Within 24 months of last patient enrolled
Time to treatment failure (TTF) | Within 24 months of last patient enrolled
Progression-free survival (PFS) using iRECIST | Within 24 months of last patient enrolled
Overall survival (OS) | Within 24 months of last patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Jose Iglesias, MD, Study Director — Consultant Chief Medical Officer for HiberCell, Inc.
Locations (7):
- United States (7):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - Sarah Cannon Research Institute /Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No